CLINICAL TRIAL: NCT04933955
Title: Comparative Evaluation of Post Operative Pain and Success Rate After Pulpotomy Using Different Tricalcium Silicate Based Materials (A Randomized Clinical Trial )
Brief Title: Evaluation of Post Operative Pain and Success Rate After Pulpotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shehab El Din Mohamed Saber, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7/6/21
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Root Canal Infection
Keywords: pulpotomy; Tricalcium silicate; Biodentine; vital pulp therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- biodentine (Active Comparator): pulptomy with biodentine
  Interventions: Procedure: vital pulp therapy
- Theracal PT (Active Comparator): pulpotomy with Theracal PT
  Interventions: Procedure: vital pulp therapy
- Neo Putty (Active Comparator): pulpotomy with Neo putty
  Interventions: Procedure: vital pulp therapy

INTERVENTIONS:
Procedure: vital pulp therapy — pulpotomy

SUMMARY:
The aim of this randomized controlled trial is to assess the post-operative pain as primary outcome and the success rate as secondary outcome after pulpotomy using different calcium silicate based materials in mature permanent teeth diagnosed with irreversible pulpitis.

DETAILED DESCRIPTION:
Setting and location :

Out-patients clinic of Endodontic Department, Faculty of Dentistry, Ain Shams University

Patient allocation:

Using computer generated randomization (www.randome.org), the participants will allocated randomly into three groups .

The sequentially numbers that will be generated, will be placed in opaque envelope until the intervention and each participant will be asked to select an envelope that determine which group of intervention he will be assigned.

Patient Classification:

Patients will be randomly divided into three groups according to material used in pulpotomy Group (1) Biodentine (n=20) Group (2) theracal PT (n=20) Group (3) Neoputty (n=20)

Procedural steps:

* Pain scale chart will be given to each patient to rate his /her pain level before endodontic treatment as preoperative reading on a visual analogue scale (VAS)
* Tooth will be anaesthetized using Local anesthesia containing Articaine with epinephrine 1:100,000.
* Rubber dam isolation of tooth
* Tooth surface disinfection using guaze soaked in 5.25% sodium hypochlorite
* Access cavity will be performed using a carbide steel round bur and tapered diamond stone until complete deroofing.
* Using a sterile excavator, the coronal pulp tissue will be excavated14
* Cotton pellets soaked in 2.5 % sodium hypochlorite will be used to achieve hemostasis for 2-3 minutes
* Once hemostasis will be achieved one of the three materials will be placed according to the manufacturer's instructions
* Final restoration will be placed

Methods of evaluation

1. Post operative pain
2. Pulpotomy success rate

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20 and 40 years old.

  * Teeth diagnosed with symptomatic irreversible pulpitis.
  * Normal periapical condition confirmed by normal periapical radiograph or that with minimal widening of the PDL space.
  * The teeth are restorable.
  * Teeth probing depth and mobility should be within normal limits.

Exclusion Criteria:

* Teeth with immature roots

  * Non restorable teeth
  * Bleeding could not be controlled after pulpotomy in 10 minutes.
  * Medically compromised patients with systemic complication that would alter the treatment.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain | pre-operative
  Each patient will be asked to fill the visual analogue scale to rate the pain level
post operative pain | 6 hours following the end of the procedure.
  Each patient will be asked to fill the visual analogue scale to rate the pain level
post operative pain | 12 hours following the end of the procedure.
  Each patient will be asked to fill the visual analogue scale to rate the pain level
post operative pain | 24 hours following the end of the procedure.
  Each patient will be asked to fill the visual analogue scale to rate the pain level
post operative pain | 48 hours following the end of the procedure.
  Each patient will be asked to fill the visual analogue scale to rate the pain level
post operative pain | 72 hours following the end of the procedure.
  Each patient will be asked to fill the visual analogue scale to rate the pain level

SECONDARY OUTCOMES:
Pulpotomy success | 3 months after the intervention
  clinical and radiographic absence of inflammation
Pulpotomy success | 6 months after the intervention
  clinical and radiographic absence of inflammation
Pulpotomy success | 9 months after the intervention
  clinical and radiographic absence of inflammation
Pulpotomy success | 12 months after the intervention
  clinical and radiographic absence of inflammation
Pulpotomy success | 18 months after the intervention
  clinical and radiographic absence of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel Rahman Hashem, phd, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haikal L, Ferraz Dos Santos B, Vu DD, Braniste M, Dabbagh B. Biodentine Pulpotomies on Permanent Traumatized Teeth with Complicated Crown Fractures. J Endod. 2020 Sep;46(9):1204-1209. doi: 10.1016/j.joen.2020.06.003. Epub 2020 Jun 15. PMID 32553879